CLINICAL TRIAL: NCT03086239
Title: An Open-Label Study on the Safety and Tolerability of Rovalpituzumab Tesirine in Japanese Patients With Advanced, Recurrent Small Cell Lung Cancer
Brief Title: A Study on the Safety and Tolerability of Rovalpituzumab Tesirine in Japanese Patients With Advanced, Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRX001-008
Record Dates: First submitted 2017-03-17; First posted 2017-03-22 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Advanced, Recurrent Small Cell Lung Cancer; Small Cell Lung Cancer; Rovalpituzumab tesirine; Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Rovalpituzumab tesirine (Experimental): Part A Dose Escalation: Rovalpituzumab tesirine intravenous (IV) (various doses and dose regimens) on Day 1 of each 6-week cycle
  Interventions: Drug: Rovalpituzumab tesirine
- Part B: Rovalpituzumab tesirine (Experimental): Part B Dose Expansion: Rovalpituzumab tesirine dosed at regimen(s) previously demonstrated in Part A to not to exceed the maximum tolerated dose (MTD).
  Interventions: Drug: Rovalpituzumab tesirine

INTERVENTIONS:
Drug: Rovalpituzumab tesirine — Intravenous

SUMMARY:
This is a Japanese, multicenter, open-label, dose-escalation study. This is the first study to assess the safety and tolerability as well as explore the pharmacokinetics, pharmacodynamics and antitumor activity of rovalpituzumab tesirine in Japanese participants with advanced small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced, recurrent small-cell lung cancer (SCLC) with documented disease progression after at least two (2) prior systemic regimens, including at least one (1) platinum-based regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic and renal function.

Exclusion Criteria:

* No prior exposure to a pyrrolobenzodiazepine (PBD)-based drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLT) | Up to 3 weeks after the initial dose of study drug (first 3 weeks of Cycle 1)
  DLTs graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Duration of response (DOR) | First dose of study drug through at least 42 days after last dose; Up to a minimum 18 weeks after participant's first dose.
  DOR is defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Objective Response Rate (ORR) | First dose of study drug through at least 42 days after last dose; Up to a minimum 18 weeks after participant's first dose.
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | First dose of study drug through long-term follow up; Up to 24 months after participant's first dose.
  OS is defined as the time from the date of first dose to the date of death.
Progression-free survival (PFS) | First dose of study drug through at least 42 days after last dose; Up to a minimum 18 weeks after participant's first dose.
  PFS time is defined as the time from the first dose of study drug to progression or death, whichever occurs first.
Clinical benefit rate (CBR) | First dose of study drug through at least 42 days after last dose; Up to a minimum 18 weeks after participant's first dose.
  CBR is defined as the proportion of participants whose overall response is either CR, PR, or Stable Disease (SD) according to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (5):
- Japan (5):
  - National Cancer Ctr Hosp East /ID# 161432, Kashiwa-shi, Chiba
  - Kyushu University Hospital /ID# 161430, Fukuoka, Fukuoka
  - Kinki University -Osakasayama Campus /ID# 161431, Osakasayama-shi, Osaka
  - National Cancer Center Hospital /ID# 161429, Chuo-ku, Tokyo
  - Wakayama Medical University /ID# 161428, Wakayama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Udagawa H, Akamatsu H, Tanaka K, Takeda M, Kanda S, Kirita K, Teraoka S, Nakagawa K, Fujiwara Y, Yasuda I, Okubo S, Shintani M, Kosloski MP, Scripture C, Tamura T, Okamoto I. Phase I safety and pharmacokinetics study of rovalpituzumab tesirine in Japanese patients with advanced, recurrent small cell lung cancer. Lung Cancer. 2019 Sep;135:145-150. doi: 10.1016/j.lungcan.2019.07.025. Epub 2019 Jul 24. PMID 31446987
- [Derived] Tanaka K, Isse K, Fujihira T, Takenoyama M, Saunders L, Bheddah S, Nakanishi Y, Okamoto I. Prevalence of Delta-like protein 3 expression in patients with small cell lung cancer. Lung Cancer. 2018 Jan;115:116-120. doi: 10.1016/j.lungcan.2017.11.018. Epub 2017 Nov 22. PMID 29290251